CLINICAL TRIAL: NCT03201848
Title: A Multisite, Randomized, Double-Blind, Placebo-Controlled, and Parallel Study to Evaluate the Efficacy and Safety of Huaiqihuang Granule in Children With Chronic Primary Immune Thrombocytopenia (Qi Yin Deficiency)
Brief Title: The Efficacy and Safety of Huaiqihuang Granule in Children With Chronic Primary Immune Thrombocytopenia
Acronym: ITP
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Qidong Gaitianli Medicines Co., Ltd (Industry)
Collaborators: Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HQH-201703.01
Record Dates: First submitted 2017-06-27; First posted 2017-06-28 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Immune Thrombocytopenia
Keywords: Huaiqihuang granule; immune thrombocytopenia; randomized; double-blind; placebo-controlled,
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — huai qi huang

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Huaiqihuang Granule (Experimental): Huaiqihuang Granule given to subject will be adjusted by body weight with treatment duration for 48 weeks
  Interventions: Drug: Huaiqihuang Granule
- Placebo (Placebo Comparator): Placebo given to subject will be adjusted by body weight After 24 weeks of placebo, change to Huaiqihuang Granule for another 24 weeks.
  Interventions: Drug: Placebo; Drug: Huaiqihuang Granule

INTERVENTIONS:
Drug: Placebo — Placebo given to subject will be adjusted by body weight (<10kg, Placebo given to subject will be adjusted by body weight(<10kg, half a bag, 2 times a day; 10-20kg; 1 bag, 2 times a day; 20-30kg, 1.5 bag, 2 times a day; 30-50kg, 2 bags, 2 times a day; ≥50kg, 3 bags, 2 times a day;) .
  Arms: Placebo
Drug: Huaiqihuang Granule — Huaiqihuang Granule given to subject will be adjusted by body weight (<10kg, half a bag, 2 times a day; 10-20kg; 1 bag, 2 times a day; 20-30kg, 1.5 bag, 2 times a day; 30-50kg, 2 bags, 2 times a day; ≥50kg, 3 bags, 2 times a day)
  Other Names: Huaiqihuang

SUMMARY:
This is a multisite, double-blind, randomized, placebo-controlled, and parallel study designed to evaluate the clinical efficacy and safety of Huaiqihuang granule for treatment to children with chronic primary immune thrombocytopenia (Qi Yin deficiency).

DETAILED DESCRIPTION:
The randomized clinical trial included subjects (n =216) will be randomly divided into experimental (n = 162) and control groups (n =54) according to a random number table. Patients in the experimental group will receive Huaiqihuang Granule . Patients in the control group will receive placebo a placebo-controlled designed is used for this study. To minimize the risks, treatment stopping rules and subsequent measures are established for subjects whose disease under study become worsening during the study. Subjects receiving placebo treatment will switch to investigational drug after Week 24 to reduce the risk of lack of efficacy by placebo.

The primary outcome measures is proportion of patients whose hemorrhage has improved (clinical effective rate).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged between 1 and 14 years (inclusive) ;
2. Is diagnosed as immune thrombocytopenia according to the criteria of ICD-10, i.e., platelet < 100×109/L for at least two hematology tests with normal blood cell morphology; skin petechia, ecchymosis and (or) the clinical manifestations of mucosa and visceral hemorrhage; no splenomegaly; exclusion of other secondary thrombocytopenia, such as aplastic leukemia, aplastic anemia characterized by thrombocytopenia as the first hematologic abnormality, hereditary thrombocytopenia, thrombocytopenia secondary to other autoimmune diseases, infections or drugs etc...
3. Meet the diagnosis criteria for Qi Yin deficiency in traditional Chinese medicine;
4. Time since initial diagnosis of ITP until randomization is at least 12 month, i.e., course of disease ≥1 year;
5. Values of prothrombin time (PT/INR) and activated partial thromboplastin time (aPTT) are within 1.2 times of normal reference range;
6. Values of biochemistry parameters including creatinine, ALT, AST, glucose, total bilirubin are less than 1.2 time of the corresponding upper limit of normal range;
7. Has signed and dated the informed consent in volunteer by the subject and the subject's legal guardian(s) (for subject who is less than 8 years old, the informed consent will be signed and dated by the subject's legal guardian(s) in volunteer).

Exclusion Criteria:

1. Is diagnosed as congenital thrombocytopenia;
2. Is diagnosed as secondary thrombocytopenia;
3. Is diagnosed as non-immune thrombocytopenia;
4. Has medical history of diabetes;
5. In the judgement of Investigator, the subject is not appropriate to participate in this study.

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 216 (Estimated)
Dates: Start 2017-11-16 (Actual); Primary Completion 2023-10-14 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
the proportion of subjects whose hemorrhage has improved (clinical effective rate) | 24、48 and 60 Weeks after treatment
  The improvement of hemorrhage is defined if at least one of the following criteria is met:
  1. Severity of hemorrhage decreases one or more grade, the severity of hemorrhage is defined as following: none: there is any hemorrhage manifestation; mild: simple (often related with an unnoticeable minor collision without obvious ecchymosis) or obvious ecchymosis by collision; moderate: mucous membrane hemorrhage (nose hemorrhage, gum, oral mucosa) and menorrhagia; and severe: organ hemorrhage (digestive tract, respiratory tract, intracranial, etc.).
  2. Significant increase in platelet count defined as platelet count is over 30×109/L and increases more than twice compared with the baseline. The results must be tested at least twice with at least 7 days apart).
  3. The score of quality of life improves one or more points.

SECONDARY OUTCOMES:
the recovery rate of immune function | 24、48 and 60 Weeks after treatment
  The recovery rate of immune function is the proportion of subjects who have normalized immune function after treatment. The parameters of immune function include cytokines, lymphocyte subsets and auto immunity. One of the three tests has been restored to normal is defined as the immune function has returned to normal.
the recovery rate of thyroid function | 12、24、36、48、60 and 72 Weeks after treatment
  The recovery rate of thyroid function is the proportion of subjects who have normalized immune function after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Runming Jin, Professor, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (14):
- China (14):
  - Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital of Tongji Medical College, Huazhong University of Science & Technology, Wuhan, Hubei
  - Wuhan Children's Hospital, Wuhan, Hubei
  - Children's Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Children's Hospital of Soochow University, Suzhou, Jiangsu
  - Jiangxi Provincial Children's Hospital, Nanchang, Jiangxi
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - The Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Beijing Children's Hospital. Capital Medical University, Beijing
  - Children's Hospital Capital Institute of Pediatrics, Beijing
  - Xinhua Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai

IPD SHARING:
Plan to Share IPD: No